CLINICAL TRIAL: NCT02949843
Title: Phase II Pilot Study Evaluating Strategies to Overcome Resistance at the Time of Progression for Patients With Non-small Cell Lung Cancers Harboring Major Oncogenic Drivers
Brief Title: Targeted Therapy in Treating Patients With Incurable Non-Small Cell Lung Cancer With Genetic Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, closed by IRB
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00041150; NCI-2016-01589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 62716 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: EGFR Activating Mutation; Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy; Adjuvants, Immunologic; Nivolumab; pembrolizumab; Molecular Targeted Therapy; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (nivolumab, pembrolizumab) (Experimental): Patients receive nivolumab IV over 60 minutes every 2 weeks or pembrolizumab IV every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: Pembrolizumab
- Arm II (kinase inhibitor, chemotherapy, immunotherapy) (Experimental): Patients receive tyrosine kinase inhibitor therapy PO targeting the initial oncogenic driver or other treatment for about 3 weeks.
  Interventions: Drug: Chemotherapy; Biological: Immunotherapy; Other: Laboratory Biomarker Analysis; Drug: Tyrosine Kinase Inhibitor
- Arm III (kinase inhibitor, targeted therapy, other treatment) (Experimental): Patients receive tyrosine kinase inhibitor therapy PO targeting initial oncogenic driver, a drug targeting the secondary mutation, or other treatment for about 3 weeks.
  Interventions: Drug: Chemotherapy; Biological: Immunotherapy; Other: Laboratory Biomarker Analysis; Drug: Targeted Molecular Therapy; Drug: Tyrosine Kinase Inhibitor

INTERVENTIONS:
Drug: Chemotherapy — Receive other treatment
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Arm II (kinase inhibitor, chemotherapy, immunotherapy); Arm III (kinase inhibitor, targeted therapy, other treatment)
Biological: Immunotherapy — Receive other treatment
  Other Names: Immunologically Directed Therapy
  Arms: Arm II (kinase inhibitor, chemotherapy, immunotherapy); Arm III (kinase inhibitor, targeted therapy, other treatment)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm I (nivolumab, pembrolizumab)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm I (nivolumab, pembrolizumab)
Drug: Targeted Molecular Therapy — Receive drug targeting secondary mutation
  Other Names: molecularly targeted therapy
  Arms: Arm III (kinase inhibitor, targeted therapy, other treatment)
Drug: Tyrosine Kinase Inhibitor — Given PO
  Other Names: Protein Tyrosine Kinase Inhibitors; PTK Inhibitors; TK Inhibitors
  Arms: Arm II (kinase inhibitor, chemotherapy, immunotherapy); Arm III (kinase inhibitor, targeted therapy, other treatment)

SUMMARY:
This phase II trial studies how well targeted therapy works in treating patients with incurable non-small cell lung cancer with a genetic mutation. Giving drugs that target other genetic mutations or other specific proteins may work better when a patient has cancer caused by a driver mutation and the treatment that targets that mutation stops working.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate among patients with high PD-L1 expressing cancers after failure of targeted therapy.

SECONDARY OBJECTIVES:

I. To compare the overall survival for patients receiving treatment targeting primary mutations, secondary mutations, or immunotherapy at the time of progression on tyrosine kinase inhibitor therapy.

II. To assess the incidence of secondary mutations in this population according to smoking status.

III. To evaluate the response rates of patients treated using these different approaches.

IV. To correlate outcomes with specific secondary genetic changes.

OUTLINE: Patients are assigned to 1 of 3 treatment arms.

ARM I (PD-L1 >= 50%): Patients receive nivolumab intravenously (IV) over 60 minutes every 2 weeks or pembrolizumab IV every 3 weeks in the absence of disease progression or unacceptable toxicity.

ARM II (PD-L1 < 50% without secondary oncogenic driver): Patients receive tyrosine kinase inhibitor therapy orally (PO) targeting the initial oncogenic driver or other treatment for about 3 weeks.

ARM III (PD-L1 < 50% with secondary oncogenic driver): Patients receive tyrosine kinase inhibitor therapy PO targeting initial oncogenic driver, a drug targeting the secondary mutation, or other treatment for about 3 weeks.

After completion of study treatment, patients are followed up for a minimum of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed incurable non-small cell lung cancer that harbors an activating mutation in EGFR, MET, BRAF, V600E, RET, HER2, translocation in Alk, or translocation in ROS-1
* Patients must be receiving treatment or planning to start treatment with a tyrosine kinase inhibitor targeting the activated gene
* Patients may not be receiving the treatment targeting the activated gene as part of a clinical treatment trial other than the Precision Oncology Trial
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine transaminase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Emergent need for palliative radiation
* Patients may not be receiving any other investigational agents for the treatment of non-small cell lung cancer
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded; breastfeeding should be discontinued

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Petty, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen patients were enrolled in the study from March 2017 to January 2018. Thirteen patients did not progress on the initial tyrosine kinase inhibitor treatment within one year. The data entered here relate to the six patients who did progress within one year.
Pre-assignment Details: Thirteen patients did not progress within one year after treatment with a tyrosine kinase inhibitor and did not continue on the study.
Period: Overall Study
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Started | 1 | 2 | 3
Completed | 1 | 1 | 2
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment) | Total
Number analyzed (Participants) | 1 | 2 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (0) | 54.5 (17.7) | 63.7 (3.5) | 60.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian (White) | 0 | 1 | 2 | 3
  Race: African American (Black) | 0 | 1 | 0 | 1
  Race: Asian | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate in Patients With High PD-L1 Expressing Cancers After Failure of Targeted Therapy Defined as Complete or Partial Response According to the Investigator's Assessment
Description: Objective Response is defined as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). This outcome applies only to Arm I. * Complete Response (CR): Disappearance of all target lesions, * Partial Response (PR): At least a 30% decrease in the sum of the target lesions Progressive Disease (PD): At least a 20% increase in the sum of the target lesions, Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease
Time Frame: Up to 1 year after failure of targeted therapy
Population: This outcome applies only to Arm I.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 1 | 0 | 0
Participants
  Partial Response | 1 | 0 | 0
  Stable Disease | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events Measured Using Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicities for each group will be estimated and described using counts and frequencies by grade, location and relatedness.
Time Frame: Adverse events were collected following each cycle of treatment (1-4) and up to 30 days after the last dose of study treatment. The average collection time from start of treatment was 7 weeks, with a range of 3 to 11 weeks.
Population: One patient in Arm II refused additional treatment and was not evaluated for adverse events, although this patient was followed for survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 1 | 1 | 3
Participants | 1 | 1 | 3

3. Secondary Outcome: Number of Mutations in Secondary Genes for Patients With PD-L1 Expression < 50%
Description: This outcome applies to only Arms II and III.
Time Frame: Up to 1 year after failure of targeted therapy
Population: This outcome applies only to Arms II and III; secondary gene mutation testing was not done in Arm I.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 0 | 2 | 3
Participants
  No secondary driver identified |  | 2 | 0
  T790M |  | 0 | 2
  Alk G1202R plus ROS-1 |  | 0 | 1

4. Secondary Outcome: Objective Response Rates for Patients Without High PD-L1 Expressing Cancers
Description: Objective response rates will be estimated in the two PD-L1 expression < 50% arms. At the time of protocol development, the intention was to estimate confidence intervals for each of these rates, and to make an exploratory comparison among the three groups comparing complete response/partial response versus stable disease/progressive disease among the groups using a Fisher's exact test (for the 2x3 table). Due to the low numbers of patients evaluable for response, these analyses were not performed.
Time Frame: Up to 3 years after failure of targeted therapy
Population: One patient in Arm II refused additional treatment and is not evaluable for response; one patient in Arm III expired one month after starting secondary treatment and is not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 1 | 1 | 2
Participants
  Partial Response | 1 | 0 | 1
  Progressive Disease | 0 | 1 | 1

5. Secondary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier methods and survival rates will be compared using log-rank tests.
  Note: Log-rank tests will not be used due to the very low sample size.
Time Frame: From date of progression on primary targeted treatment to death, assessed up to 3 years.
Population: Patient records were reviewed at this time for all six patients.
Measure: Median (Full Range); unit: months
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 1 | 2 | 3
months | 36 [36 to 36] | 8.3 [0.72 to 15.94] | 2.56 [1.08 to 36]

6. Secondary Outcome: Rate of Tobacco Use and Mutation Burden Based on PD-L1 Expression at Time of Progression
Description: Smoking History was defined as Never, Former or Current
Time Frame: Assessed at enrollment into study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
Number analyzed (Participants) | 1 | 2 | 3
Participants
  Never Smoked | 1 | 2 | 1
  Formerly Smoked | 0 | 0 | 2
  Currently Smoke | 0 | 0 | 0
Statistical Analysis 1: Comparison: Arm I (Nivolumab, Pembrolizumab) vs Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) vs Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment); Null Hypothesis is that each arm has equal rates of smoking history; Test type: Other; p = 0.6, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected following each cycle of treatment (1-4), and up to 30 days following the last dose of study treatment. The average collection time from start of treatment was 7 weeks, with a range of 3 to 11 weeks. One patient refused additional treatment after the initial progression and was not followed for adverse events, but was followed for mortality.
Arm/Group | Arm I (Nivolumab, Pembrolizumab) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment)
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nivolumab, Pembrolizumab) (N=1) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) (N=1) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment) (N=3)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Nivolumab, Pembrolizumab) (N=1) | Arm II (Kinase Inhibitor, Chemotherapy, Immunotherapy) (N=1) | Arm III (Kinase Inhibitor, Targeted Therapy, Other Treatment) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 2 (4)
Leukocytotsis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (3) | 1 (1) | 3 (5)
Fatigue (General disorders) | 1 (2) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (4) | 1 (1) | 3 (5)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (1) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 1 (1) | 3 (5)
Creatinine increased (Investigations) | 1 (4) | 0 (0) | 3 (5)
Platelet count decreased (Investigations) | 1 (4) | 1 (1) | 3 (5)
White blood cell decreased (Investigations) | 1 (4) | 1 (1) | 3 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 2 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02949843/Prot_SAP_001.pdf
  • Informed Consent Form (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT02949843/ICF_000.pdf